CLINICAL TRIAL: NCT01543009
Title: Use of Local Warming in Children to Facilitate Venipuncture. A Randomized Controlled Trial.
Brief Title: Use of Local Warming in Children Venipuncture
Status: Suspended | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulty in recruiting
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Filippo Festini, Professor of Nursing, University of Florence
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UFI2012WARM
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Phobia Phlebotomy
Keywords: child; venipuncture; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emla + no additional intervention (No Intervention): Children in this arm will receive standard preparation of the venipuncture site (local analgesia with Emla) without warming
- Emla + Local Warming (Experimental): Children in this arm will receive standard preparation of the venipuncture site (local analgesia with Emla) plus warming with a heating pad at 40°C for 5 minutes
  Interventions: Other: Emla + Local Warming

INTERVENTIONS:
Other: Emla + Local Warming — In this arm Emla is applied 60 minutes before the procedure and then the site of venepuncture is warmed by an electric heating sand pad at the temperature of 40°C for 5 minutes before performing cannulation
  Arms: Emla + Local Warming

SUMMARY:
The aim of this study is to determine if local application of heat increases the probability of insertion of peripheral venous catheter at the first attempt, reduces the time needed to obtain cannulation and maintains the analgesic effect of Emla in children undergoing peripheral venous cannulation and previously treated with local analgesia with Emla.

ELIGIBILITY:
Inclusion Criteria:

* age between 8 and 13 years
* Intravenous drug therapy prescribed by a physician
* no allergy to lidocaine
* no local skin disease
* absence of burns scars
* child and his/her family are native speaker of Italian
* BMI not lower than 10° centile for sex and age according to the CDC standards

Exclusion Criteria:

* age of child not included in the age range established for the study
* Intravenous drug therapy not needed
* Presence of an allergy to lidocaine products
* Skin disease
* Presence of burns scars
* The child or his/her family are not native speaker Italian
* BMI lower than 10° centile according to the CDC standards

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
rate of success of peripheral venous cannulation at the first attempt | The outcome is observed and recorded immediatly after the venous cannulation. No follow up is required

SECONDARY OUTCOMES:
pain perceived by the child undergone to the cannulation | The outcome is observed and recorded immediatly after the venous cannulation. No follow up is required
  The pain level is estimated using a visual analog scale (from 0 to 10) or the Wong "faces'" Scale
Difficulty in performing cannulation perceived by Nurse | The outcome is observed and recorded immediatly after the venous cannulation. No follow up is required
  This outcome is calculated using an "ad hoc" Visual Analog Scale (from 0 to 10)
Time needed to obtain cannulation | From positioning tourniquet to completion of cannulation. No follow up is required
  Time is calculated in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Festini, RN, BA, BSN, MSN, Principal Investigator — University of Florence
Locations (1):
- Meyer Children Hospital, Florence, Italy